CLINICAL TRIAL: NCT00627614
Title: Identification and Differentiation of Breast Masses by Vibro-Acoustography
Brief Title: Vibro-Acoustography Imaging in Diagnosing Breast Masses in Women With a Breast Mass or Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Azra Alizad, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 284-06; P30CA015083 (NIH); CDR0000583016 (Other: NCI)
Record Dates: First submitted 2008-02-29; First posted 2008-03-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- breast imaging study (Experimental)
  Interventions: Other: breast imaging study

INTERVENTIONS:
Other: breast imaging study — 1. A set of vibro-acoustography (VA) scans will be taken of the breast by an experimental vibro-acoustography device that uses ultrasound for imaging.
  2- An ultrasound scan (sonography) of the breast using a clinical ultrasound machine may be taken during the procedure.

SUMMARY:
RATIONALE: New diagnostic procedures, such as vibro-acoustography imaging, may be an effective method of diagnosing breast cancer.

PURPOSE: This clinical trial is studying how well vibro-acoustography imaging works in diagnosing breast masses in women with a breast mass or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To study in vivo detection of breast masses by vibro-acoustography (VA) imaging.
* To evaluate the performance of VA imaging in differentiating between benign and malignant breast masses identified as BI-RADS 4 or 5.

OUTLINE: Patients undergo clinical mammography of the breast, followed by vibro-acoustography (VA) imaging using ultrasonography over 90 minutes. Patients may also undergo further imaging using clinical ultrasonography.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspiciuos breast lesions identified as BI-RADS 4 or 5 and 3
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Not pregnant
* No condition that does not allow proper use of study imaging devices

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Detection and differentiation of breast masses with an estimated specificity of ≥ 70% using vibro-acoustography (VA) imaging | 25 minutes for Breast VA imaging

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

REFERENCES:
- [Result] Alizad A, Whaley DH, Urban MW, Carter RE, Kinnick RR, Greenleaf JF, Fatemi M. Breast vibro-acoustography: initial results show promise. Breast Cancer Res. 2012 Sep 29;14(5):R128. doi: 10.1186/bcr3323. PMID 23021305
- [Result] Urban MW, Chalek C, Haider B, Thomenius KE, Fatemi M, Alizad A. A beamforming study for implementation of vibro-acoustography with a 1.75-D array transducer. IEEE Trans Ultrason Ferroelectr Freq Control. 2013 Mar;60(3):535-51. doi: 10.1109/TUFFC.2013.2595. PMID 23475919
- [Result] Kamimura HA, Urban MW, Carneiro AA, Fatemi M, Alizad A. Vibro-acoustography beam formation with reconfigurable arrays. IEEE Trans Ultrason Ferroelectr Freq Control. 2012 Jul;59(7):1421-31. doi: 10.1109/TUFFC.2012.2343. PMID 22828838
- [Result] Urban MW, Alizad A, Aquino W, Greenleaf JF, Fatemi M. A Review of Vibro-acoustography and its Applications in Medicine. Curr Med Imaging Rev. 2011 Nov 1;7(4):350-359. doi: 10.2174/157340511798038648. PMID 22423235
- [Result] Chen S, Aquino W, Alizad A, Urban MW, Kinnick R, Greenleaf JF, Fatemi M. Thermal safety of vibro-acoustography using a confocal transducer. Ultrasound Med Biol. 2010 Feb;36(2):343-9. doi: 10.1016/j.ultrasmedbio.2009.10.003. PMID 20113864
- [Result] Alizad A, Whaley DH, Greenleaf JF, Fatemi M. Image features in medical vibro-acoustography: in vitro and in vivo results. Ultrasonics. 2008 Nov;48(6-7):559-62. doi: 10.1016/j.ultras.2008.04.014. Epub 2008 May 25. PMID 18599102